CLINICAL TRIAL: NCT04597463
Title: The Combination of Endometrial Injury and Freeze All Strategy in Women With a History of Repeated Implantation Failure.
Brief Title: The Combination of Endometrial Injury and Freeze All Strategy in Women With a History of RIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, IOANNIS RIGOS, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1811198218111982
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Endometrial Injury; Hysteroscopy; Repeated Implantation Failures
Keywords: Endometrial injury; Hysteroscopy; RIF; IVF; ART

STUDY DESIGN:
Intervention Model Description: Endometrial injury in RIF patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endometrial injury (Experimental): Endometrial injury before the embryo transfer of a frozen cycle
  Interventions: Procedure: Endometrial injury

INTERVENTIONS:
Procedure: Endometrial injury — Endometrial injury was performed hysteroscopically after freeze all cycles and during the cycle before the frozen embryo transfer

SUMMARY:
The investigators checked the hypothesis whether endometrial injury performed during the cycle before a frozen embryo transfer in women with RIF can improve pregnancy rates

DETAILED DESCRIPTION:
After a freeze all cycle, participants were divided in two groups: an intervention group (n=30), who underwent endometrial injury before the transfer, and a control group (n=30), who underwent no other intervention. The primary outcome was clinical pregnancy rate, while secondary clinical and laboratory parameters. Baseline and cycle characteristics were also compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with RIF under 42 years old
* BMI 20-30
* Normal endometrial cavity
* FSH <15 IU/L
* Absence of immunological or hematological disorder

Exclusion Criteria:

* women over 42 years old
* FSH>15 IU/L
* women with chronic immunological or hematological disorder
* stage III or IV of endometriosis
* women with pathology concerning the endometrial cavity
* women with a medical history of adnexectomy or oophorectomy

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Physiological parameter - Live birth rate | 22 weeks
  The complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age

SECONDARY OUTCOMES:
Physiological parameter -Clinical pregnancy rate | 7 weeks
  A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy
Adverse event - Miscarriage | 22 weeks
  Spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Siristatidis, Prof, Study Director — National and Kapodistrian University of Athens
Locations (1):
- National and Kapodistrian University of Athens, Athens, Greece

REFERENCES:
- [Background] Basile N, Garcia-Velasco JA. The state of "freeze-for-all" in human ARTs. J Assist Reprod Genet. 2016 Dec;33(12):1543-1550. doi: 10.1007/s10815-016-0799-9. Epub 2016 Sep 14. PMID 27629122
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Background] Wong KM, van Wely M, Mol F, Repping S, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2017 Mar 28;3(3):CD011184. doi: 10.1002/14651858.CD011184.pub2. PMID 28349510